CLINICAL TRIAL: NCT05753514
Title: Radial Extracorporeal Shockwave Therapy (rESWT) for Coccydynia: a Quasi-experimental Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Kabir Singh Lota, Doctor, Barts & The London NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-09
Record Dates: First submitted 2023-02-12; First posted 2023-03-03 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Coccyx Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESWT (Experimental): Effect of ESWT in alleviating pain
  Interventions: Other: ESWT

INTERVENTIONS:
Other: ESWT — ESWT

SUMMARY:
The aim of this study was to assess whether a pain-adapted protocol of rESWT is effective in treating coccydynia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* VAS pain level ≥6
* Diagnosis of coccydynia (persistent pain in the coccygeal area consistent with coccydynia)

Exclusion Criteria:

* Age <18 years
* Local or systemic neurological disease
* Rheumatological disease
* Malignant disease
* Previous spinal surgery or spinal disease
* Coagulopathies
* Pregnancy
* VAS pain level <6
* Recent (≤6 weeks) trauma to the coccyx

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Management of coccydynia | 12 months
  Management of coccydynia (pain in the coccyx). The main presenting symptom is pain. its management is the primary goal of treatment. The pain VAS was used to monitor patient response and clinical improvement throughout treatment, with patients ranking the severity of their pain at rest, between "no pain" (0) and "worst imaginable pain" (10). Patients were asked their pain level before treatment at each session; although, this did not form part of our formal data collection. Treatment continued until patients reported a VAS pain level ≤3, at which point they were discharged from the clinic.

IPD SHARING:
Plan to Share IPD: Yes